CLINICAL TRIAL: NCT06536400
Title: A Phase I, Open-label, Dose-escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic of HSK42360 in Patients With BRAF V600 Mutation Locally Advanced or Metastatic Solid Tumors
Brief Title: Phase I Study of HSK42360 in Solid Tumors With BRAF V600 Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSK42360-101
Record Dates: First submitted 2024-07-24; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase Ia (Part A): HSK42360 as monotherapy (Experimental): Phase 1a (Part A): dose escalation of HSK42360 as monotherapy at various dose levels
  Interventions: Drug: HSK42360
- Phase Ia (Part B): HSK42360 as monotherapy (Experimental): Phase 1a (Part B): dose extention of HSK42360 as monotherapy at certain dose levels
  Interventions: Drug: HSK42360
- Phase Ib: HSK42360 as monotherapy (Experimental): Phase 1b: dose expansion for HSK40118 as monotherapy at a dose determined during Phase 1a (Part B) in patients with BRAF V600 mutation locally advanced or metastatic solid tumors
  Interventions: Drug: HSK42360

INTERVENTIONS:
Drug: HSK42360 — Oral administration, QD

SUMMARY:
This is a phase I, open-label, dose-escalation and expansion study to evaluate the safety, tolerability, PK and PD of HSK42360 when given orally in patients with active BRAF V600 mutation locally advanced or metastatic Solid Tumors.

DETAILED DESCRIPTION:
The study will contain two phases: Phase Ia is dose escalation phase and Phase Ib is dose expansion phase.

Phase Ia will contain two part: Dose Escalation Part (Part A) and Extension Part (Part B). Part A based on the "3+3" design for dose escalation and safety evaluation requirements. Patient cohorts at selected doses may be extended to further investigate the tolerability, PK and PD of HSK42360. The number of patients to be enrolled will be up to 10 subjects in each Part B cohort. Approximately 30-70 subjects will be enrolled in Phase Ia.

Phase Ib no less than 10-50 subjects will be enrolled in each expansion cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years，Male and female patients, at time of signing informed consent form (ICF).
2. ECOG performance status 0-1, or KPS (Karnofsky Performance Status) Score>60.
3. Life expectancy ≥ 3 months.
4. Patients with locally advanced or metastatic solid tumors confirmed by histology or cytology, who have failed standard treatment (disease progression after treatment or intolerable treatment); patients who have previously received BRAF and/or MEK inhibitor therapy are allowed to be included in this study.
5. Positive BRAF V600 mutation result confirmed prior to the administration of HSK42360.
6. Patients will provide blood or tumor sample according to their own willingness.
7. Measurable or non-measurable disease by RECIST 1.1 or RANO criteria.
8. Brain metastasis patients with inactive CNS lesions; Original intracranial tumor patient with inactive CNS lesions, or patients treated with ≤4mg/day corticosteroid and without convulsion for ≥2 weeks.
9. Adequate hematologic, hepatic, and renal function.
10. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days after the last dose.

Exclusion Criteria:

1. malignant tumor within 2 years, with the exception of cutaneous squamous cell carcinoma, cervical carcinoma in situ, papillary thyroid carcinoma, or other tumors with low malignancy.
2. Uncontrollable pleural effusion, ascites, or pericardial effusion per protocol.
3. Treatment with any of the following:

   Prior treatment with anti-tumor drug within 4 weeks or approximately 5 × t1/2 prior to the first dose of HSK42360, whichever is shorter; Prior treatment with nitrosourea or mitomycin C within 6 weeks prior to the first dose of HSK42360; Prior treatment with palliative radiotherapy or anti-tumor herbs within 2 weeks prior to the first dose of HSK42360; Prior treatment with radiotherapy, electric field therapy, or other anti-tumor therapies within 4 weeks prior to the first dose of HSK42360.
4. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment, with the exception of alopecia, dermal toxicity, and other toxicity considering no safety risks by investigator.
5. Any disease which would preclude drug absorption, metabolism or pharmacokinetics, e.g. active peptic ulcer or chronic gastroesophageal reflux disease.
6. Patients who have clinically significant or uncontrolled cardiac disease, include: QTc interval ≥ 450(male)/470(female) msec; any clinically significant arrhythmia; left ventricular ejection fraction < 50%; myocardial infarction, unstable angina, or class III/IV cardiac failure by the NYHA that occurred within 6 months prior to the first dose of HSK42360.
7. Any thromboembolic events within 6 months prior to the first dose of HSK42360; any familial or acquired thrombophilia.
8. Uncontrolled hypertension (systolic pressure≥160mmHg, or diastolic pressure≥100mmHg), diabetes (fasting blood-glucose≥10mmol/L), seizures, chronic obstructive pulmonary disease (COPD), interstitial pneumonia, pulmonary interstitial fibrosis, Parkinson's disease, active bleeding, or systemic active infection.
9. Any unstable systemic disease, e.g. severe metabolic disease: liver cirrhosis, renal failure, or uremia.
10. Treatment with inhibitors/inducers for CYP3A4, or substrates of CYP3A4, CYP2C9, CYP2C8, OATP1B1, OATP1B3, OAT1, OAT3, P-gp or BCRP within 14 days or approximately 5 × t1/2 prior to the first dose of HSK42360, whichever is shorter.
11. Patient with cognitive dysfunction, or history of mental illness, other uncontrolled comorbidities, alcohol dependence, hormone dependence or drug abuse.
12. Autologous transplantation surgery within 3 months prior to the first dose of HSK42360; Allogeneic transplantation, or stem-cell Transplant surgery within 6 months prior to the first dose of HSK42360; Major surgery or significant traumatic injury occurring within 4 weeks prior to the first dose of HSK42360.
13. Patient with a history of immunodeficiency, including HIV positive, or other acquired/congenital immunodeficiency diseases.
14. Any disease of the eyes > CTCAE v5.0 Grade 1.
15. Patient with active hepatitis B or hepatitis C.
16. Patient with active syphilis infection.
17. Allergic to any HSK42360 active constituent or ingredients.
18. Participate in other clinical trials within 4 weeks prior to the first dose of HSK42360.
19. Positive pregnancy test, or breastfeeding.
20. Any other circumstances that would, in the investigator's judgment, prevent the subject's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2026-08-30 (Estimated); Study Completion 2027-07-07 (Estimated)

PRIMARY OUTCOMES:
MTD | Up to approximately 52 months
  MTD determination: dose limiting toxicity (DLT) rate
DLTs | Up to approximately 52 months
  Incidence of dose-limiting toxicities (DLTs) at Cycle 0 and Cycle1
AEs | Up to approximately 52 months
  Rate and severity of adverse events of HSK42360 as monotherapy
RP2D | Up to approximately 52 months
  RP2D determination: DLT, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary safety and anticancer activity data
ECOG Performance Status Scale | Up to approximately 52 months
  Change of the grade as a part of HSK43260 safety data
Karnofsky Performance Scale, KPS | Up to approximately 52 months
  Change of the grade as a part of HSK43260 safety data

SECONDARY OUTCOMES:
Overall response rate (ORR) | Up to approximately 52 months
  ORR, defined as the proportion of patients who experience a best response of confirmed CR or PR according to RECIST 1.1/RANO
Disease control rate (DCR) | Up to approximately 52 months
  DCR, defined as the proportion of patients who experience a best response of CR, PR, or stable disease (SD) according to RECIST 1.1
Duration of response (DOR) | Up to approximately 52 months
  DOR, defined as the time from first documented response of complete response (CR) or partial response (PR) to the date of first documented progressive disease or death due to any cause, whichever occurs first
Progression free survival (PFS) | Up to approximately 52 months
  PFS, defined as the time frocease or death due to any cause, whichever occurs first
Overall survival (OS) | Up to approximately 52 months
  OS, defined as the time from the first dose of HSK42360 until the date of death due to any cause
Area under the curve (AUC) of HSK42360 | Circle 0 (single-dose circle, 3 days) and circle 1 (multiple-dose circle, 21days)
maximum plasma concentration (Cmax) of HSK42360 | Circle 0 (single-dose circle, 3 days) and circle 1 (multiple-dose circle, 21days)
half-life (t1/2) of HSK42360 | Circle 0 (single-dose circle, 3 days) and circle 1 (multiple-dose circle, 21days)
Tmax(Time to maximum plasma concentration) of HSK42360 | Circle 0 (single-dose circle, 3 days) and circle 1 (multiple-dose circle, 21days)

OTHER OUTCOMES:
circulating tumor DNA (ctDNA) | Up to approximately 52 months
  Assess treatment-induced modulation of MAPK pathway biomarkers
phosphorylate ERK (pERK) | Up to approximately 52 months
  Assess the degradation of pERK protein

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing TianTan Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital, Nanning, Guangxi
  - The Third People's Hospital of Zhengzhou, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Hangzhou First People's Hospital, School of Medicine, Westlake University, Hangzhou, Zhejiang